CLINICAL TRIAL: NCT02485262
Title: Outcome of New Direct Acting Agents For Hepatitis C
Brief Title: Outcome of New Direct Acting Agents For Hepatitis C A Community Based Experience
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Arrowhead Regional Medical Center (Other)
Responsible Party: Principal Investigator, Zeid Kayali, MD, MD,MBA, Arrowhead Regional Medical Center
Other Study IDs: 1234; 14-25 (Other: 14-25)
Record Dates: First submitted 2015-06-19; First posted 2015-06-30 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Hepatitis C
Keywords: Protease inhibitor treatment
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir; Simeprevir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sofosbuvir and simeprevir — Hepatitis C treatment using Direct Acting Agents
  Other Names: Sovaldi and Olysio

SUMMARY:
Chronic Hepatitis C virus (HCV) infection is the leading cause of advanced liver disease worldwide. The virus successfully evades host immune detection and has highly restricted requirements for growth in vitro that for many years hampered efforts to find a safe, uncomplicated, and reliable oral antiviral therapy. Ten years after discovery, pegylated interferon-alpha and ribavirin (PR) treatment for 24-48 weeks became the standard of care (1-5). PR therapy offered limited performance and availability across the diverse spectrum of HCV disease and was fraught with excessive and often limiting side effects. The first direct acting agents (DAAs) were protease inhibitors (PIs) that were introduced in 2011 and could only be used only in combination with PR because of concerns for rapid PI viral resistance. Although the first generation PIs added increased efficacy to the PR regimen, they also added new side effects and untoward drug interactions (6-8). Sofosbuvir (SOF) is a potent nucleoside inhibitor (NI) that has recently been approved for treatment of HCV. The drug has low toxicity, high resistance barrier, and minimal drug interactions with other HCV DAAs such as PIs and anti-NS5A agents. SOF is safe and effective across different viral genotypes, disease stages, and special patient groups such as those co-infected with HIV. When used in combination with ribavirin or another DAA, SOF has revolutionized the HCV treatment spectrum and set the stage for nearly universal HCV antiviral therapy. Sustained virologic response (SVR12) for SOF plus ribavirin and pegylated interferon (PR) is 90% for genotype 1 and 85-94% for genotypes 2 and 3 (9-16). SOF plus simeprevir (protease inhibitor) showed a 94% SVR12 for genotype 1 (9-16). More so than any other anti-HCV drug developed to date, SOF offers the widest applicability for all infected patients yet can be given in a personalized regimen to maximize performance

DETAILED DESCRIPTION:
SOF plus simeprevir or PR became the backbone of HCV treatment. The demographics and characteristics of HCV patients in the Inland Empire are different than the cohort enrolled in SOF trials. There is a need to determine if the community based outcomes at match the outcome reported in the clinical trials.

Aim of the study

To propectively evaluate the efficacy and tolerability of the SOF treatment regimens prescribed at the ARMC and compare them to outcomes reported in the clinical trials that were the basis for FDA approval.

Study Description

This is a prospective registry study conducted at the ARMC. Targeted subjects are HCV patients are ARMC who received one of the SOF based treatment regimens from December 20, 2013 to December 19, 2014.

Primary end Point is sustained virological response at 12 weeks (SVR 12) and secondary end point is compliance and safety. Safety and compliance will be determined based on symptoms reported during clinic visits and number of refills and doses dispensed for every patient.

ELIGIBILITY:
Inclusion Criteria:

* Adult Chronic HCV patients aged >18
* Treatment naïve
* Patient with cirrhosis and no cirrhosis. Cirrhosis defined as stage 4 fibrosis on liver biopsy or Fibro sure results indicating cirrhosis or has clinical findings suggestive of cirrhosis
* Patients meet the indication to receive one of the SOF treatment based regimens

Exclusion Criteria:

* Co-infected patients with HIV or Hepatitis B
* Patient received one of the DAAs regimens
* Patient with active substance abuse and alcohol abuse
* Patient received prior DAA regimen
* Decompensated cirrhotic patients
* Patient has contraindication to receive SOF

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Targeted subjects are HCV patients are ARMC who received one of the SOF based treatment regimens from December 20, 2013 to May 2015
Sampling Method: Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
SVR 12 | 12 weeks post treatment

SECONDARY OUTCOMES:
Safety and Tolerability as measured by the number of participants with AEs, Change in baseline laboratory results | 24 weeks
  Number of participants with AEs, Change in baseline laboratory results

CONTACTS AND LOCATIONS:
Overall Officials: Zeid Kayali, MD,MBA, Principal Investigator — Arrowhead Regional Medical Center
Locations (1):
- Arrowhead Regional Medical Center, Colton, California, United States

REFERENCES:
- [Result] Lawitz E, Poordad FF, Pang PS, Hyland RH, Ding X, Mo H, Symonds WT, McHutchison JG, Membreno FE. Sofosbuvir and ledipasvir fixed-dose combination with and without ribavirin in treatment-naive and previously treated patients with genotype 1 hepatitis C virus infection (LONESTAR): an open-label, randomised, phase 2 trial. Lancet. 2014 Feb 8;383(9916):515-23. doi: 10.1016/S0140-6736(13)62121-2. Epub 2013 Nov 5. PMID 24209977
- [Result] Gane EJ, Roberts SK, Stedman CA, Angus PW, Ritchie B, Elston R, Ipe D, Morcos PN, Baher L, Najera I, Chu T, Lopatin U, Berrey MM, Bradford W, Laughlin M, Shulman NS, Smith PF. Oral combination therapy with a nucleoside polymerase inhibitor (RG7128) and danoprevir for chronic hepatitis C genotype 1 infection (INFORM-1): a randomised, double-blind, placebo-controlled, dose-escalation trial. Lancet. 2010 Oct 30;376(9751):1467-75. doi: 10.1016/S0140-6736(10)61384-0. Epub 2010 Oct 14. PMID 20951424
- [Result] Lawitz E, Mangia A, Wyles D, Rodriguez-Torres M, Hassanein T, Gordon SC, Schultz M, Davis MN, Kayali Z, Reddy KR, Jacobson IM, Kowdley KV, Nyberg L, Subramanian GM, Hyland RH, Arterburn S, Jiang D, McNally J, Brainard D, Symonds WT, McHutchison JG, Sheikh AM, Younossi Z, Gane EJ. Sofosbuvir for previously untreated chronic hepatitis C infection. N Engl J Med. 2013 May 16;368(20):1878-87. doi: 10.1056/NEJMoa1214853. Epub 2013 Apr 23. PMID 23607594